CLINICAL TRIAL: NCT05415163
Title: Effect of Vascular Photobiomodulation on Sleep Quality, Relaxation and Stress Control: Randomized Controlled Clinical Trial
Brief Title: Vascular Photobiomodulation on Sleep Qualityand Stress
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Lara Jansiski Motta, PhD, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PMBQS
Record Dates: First submitted 2022-06-08; First posted 2022-06-10 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Stress Disorder; Sleep Disorder
Keywords: stress; sleep disorder; photobiomodulation; laser therapy
MeSH Terms: conditions — Stress Disorders, Traumatic; Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The photobiomodulation application devices are identical in both groups and in the placebo group the device will not emit light, only the sound signal. Both participant and researcher will wear protective eyewear and will not know which equipment is the active or placebo. Only a researcher external to the procedure will know which equipment is in each group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vascular photobiomodulation (Experimental): Laser will be applied with the spot located in the radial artery of the participant's arm (right or left), and fixed to the wrist with a specific bracelet.
  Interventions: Procedure: vascular photobiomodulation
- photbiomodulation-sham (Sham Comparator): The device will be placed with the spot located in the radial artery of the participant's arm (right or left), and fixed to the wrist with a specific bracelet no laser apllied.
  Interventions: Procedure: vascular photobiomodulation

INTERVENTIONS:
Procedure: vascular photobiomodulation — application of photobiomodulation with the device O Ecco ILIB (Eccofibras, São Paulo, Brazil) containing its red wavelength 660 nm ± 10 nm and power 100 mW, with an application time of 30 minutes. The device will be positioned with the spot located in the radial artery of the participant's arm (right or left), and fixed to the wrist with a specific bracelet.

SUMMARY:
Randomized clinical trial to evaluate the effect of vascular photobiomodulation on sleep quality, relaxation and stress when compared to placebo.

DETAILED DESCRIPTION:
The quality of sleep is directly linked to the quality of human life. Irradiation of blood in the transcutaneous vascular technique is believed to decrease blood viscosity and platelet aggregation; activates superoxide dismutase; promotes increased oxygen content and stimulates microcirculation, it also stimulates increased serotonin production and cortisol reduction. Serotonin functions include sleep initiation, mood improvement, anxiety and depression. Therefore, the objective of the present project is to evaluate the effect of ILIB on salivary biomarkers related to stress and sleep. Therefore, participants with problems related to sleep quality will be selected and divided into 2 groups, group 1 undergoing ILIB Therapy twice a week for 30 minutes and group 2 the same frequency and time of application, but with placebo equipment. At the end of 10 sessions, salivary biomarkers related to stress and sleep and the patients' perception will be evaluated through specific questionnaires on the effect of ILIB on sleep, stress and relaxation.

ELIGIBILITY:
Inclusion Criteria:

* poor sleep quality.
* Participants who for at least six months have had poor sleep quality (score > 5 points), measured using the PSQI,

Exclusion Criteria:

* use medications or perform treatments that may affect the sleep cycle
* treatment for hypertension
* asthma,
* attention deficit disorder,
* diabetes.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-11-10 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Quality of sleep | five weeks
  Quality of sleep evaluated by Pittsburgh Sleep Quality Index

CONTACTS AND LOCATIONS:
Locations (1):
- Lara Motta, São Roque, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No